CLINICAL TRIAL: NCT01525719
Title: A Phase II Single Arm Study to Evaluate the Safety and Efficacy of RAD001 as Monotherapy in Treatment naïve Advanced Cholangiocarcinoma
Brief Title: Single Arm Study of RAD001 as Monotherapy in Treatment in Advanced Cholangiocarcinoma
Acronym: CRAD001T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ratchavithi Hospital (Other Government)
Responsible Party: Principal Investigator, Kawin Leelawat, Department of Surgery, Ratchavithi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-53326
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Cholangiocarcinoma
Keywords: cholangiocarcinoma; RAD001; everolimus
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10 mg everolimus
  Other Names: RAD001

SUMMARY:
The purpose of this study is to determine whether everolimus is effective in the treatment of patients with advance cholangiocarcinoma.

DETAILED DESCRIPTION:
Cholangiocarcinoma is one of the most common cause of cancer death in Thailand. Patients with cholangiocarcinoma are often diagnosed at advanced stage. Palliative therapeutic approaches consisting of percutaneous and endoscopic biliary drainage have usually been used for these patients, since there is no effective chemotherapeutic treatment for this type of cancer. Activation of the phosphoinositide-3-kinase (PI3K)/Akt/mTOR signaling pathway is frequently found in cholangiocarcinoma cells. It has been suggested to be a key step leading to the progression of cholangiocarcinoma. In this study, the investigators hypothesize that inhibition of mTOR may be useful in treating cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmed diagnosis of cholangiocarcinoma.
* Patients must present with disease not amenable to curative surgery.
* ECOG performance status of < 2
* Patients with at least one measurable lesion at baseline as per the RECIST criteria.
* The following laboratory parameters at screening (visit 1):

WBC are equal to or more than 3,000/uL. Platelet are equal to or more than 100,000/uL Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN. Patients with known liver metastases: AST and ALT ≤ 5 x ULN Total Bilirubin < 2 mg/dl* (after drainage) Serum creatinine equal to or less than 2.0 x upper normal limit

* Life expectancy equal to or more than 12 weeks.
* Ability to understand and willingness to sign a written informed consent and to be able to follow the visit schedule.
* Female patients at child-bearing age must have negative pregnancy test.
* Patients refuse to have treatment with Chemotherapy or Radiation.

Exclusion Criteria:

* Patients within 2 weeks post-minor surgery, 4 weeks post-major surgery to avoid wound healing complications. Percutaneous biopsies require no waiting time prior to study entry.
* Patients with a recent history of hemoptysis, ≥ 0.5 teaspoon of red blood.
* Patients who have received prior systemic treatment for their metastatic cholangiocarcinoma.
* Presence of clinically relevant ascites or liver failure.
* Patients with extensive symptomatic fibrosis of the lungs.
* Patients with a known hypersensitivity to RAD001 (everolimus).
* Patients who have previously received mTOR inhibitors (sirolimus, temsirolimus, everolimus, deforolimus).
* History or clinical evidence of central nervous system (CNS) metastases. Note: Subjects who have previously-treated CNS metastases (surgery±radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible:

Are asymptomatic Have had no evidence of active CNS metastases for ≥ 6 months prior to enrollment and Have no requirement for steroids or enzyme-inducing anticonvulsants (EIAC)

* Clinically significant gastrointestinal abnormalities including, but not limited to:

Malabsorption syndrome Major resection of the stomach or small bowel that could affect the absorption of RAD001 Active peptic ulcer disease Inflammatory bowel disease Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning of study treatment;

* Patients receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent. Inhaled and topical steroids are acceptable
* Patients with a known history of human immunodeficiency virus seropositivity
* Patients with autoimmune hepatitis
* Patients with an active, bleeding diathesis. Patients may use coumadin or heparin preparations.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Patients who have a history of another primary malignancy ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of uterine.
* Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods.
* Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study treatment start.
* Patients unwilling or unable to comply with the protocol.
* Patient who will have got benefit from Radiation or Chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival in cholangiocarcinoma patients whom treated with everolimus | One year

SECONDARY OUTCOMES:
overall survival rate | Two years
  Overall survival is defined as the time from dater of start of treatment to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kawin Leelawat, MD, PhD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand